CLINICAL TRIAL: NCT03182296
Title: Visualizing Beta Cells in Patients With a History of Gestational Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NL56938.091.16
Record Dates: First submitted 2017-05-29; First posted 2017-06-09 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Gestational Diabetes
Keywords: beta cell mass; exendin; GLP-1 PET
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: Comparison of women with and without a history of gestational diabetes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gestational diabetes (Experimental): Women with a history of gestational diabetes
  Interventions: Radiation: 68Ga-NODAGA-exendin-4 PET/CT
- Control (Active Comparator): Women without a history of gestational diabetes
  Interventions: Radiation: 68Ga-NODAGA-exendin-4 PET/CT

INTERVENTIONS:
Radiation: 68Ga-NODAGA-exendin-4 PET/CT — 68Ga-NODAGA-exendin-4 PET/CT

SUMMARY:
In order to evaluate the difference in beta cell mass in women with and without a history of gestational diabetes mellitus (GDM), investigators aim to compare quantitative PET imaging of the pancreas between these groups. Investigators propose to measure uptake of 68Ga-NODAGA-exendin-4 in the pancreatic beta cells of these women as a measure for beta cell mass. Furthermore, investigators aim to compare uptake of the radiolabeled tracer to beta cell function measured by laboratory parameters. These highly relevant data within this at-risk population for type 2 diabetes (T2D) will provide the investigators with more information on the role of beta cell mass in the predisposition for development of T2D leading to better knowledge on the pathophysiology of this disease. This could be of great interest for development of new treatment options.

DETAILED DESCRIPTION:
Gestational diabetes Insulin is produced by pancreatic beta cells and is needed for optimal glucose homeostasis. In healthy individuals, the mass and function of beta cells changes to adapt to variations in insulin demand in the body. For example, adaptive beta cell hyperplasia, hypertrophy and hyperfunction occur in situations of increased metabolic demand, like pregnancy.

In rodents a 2-3 fold increase in beta cell mass is observed at the end of gestation. By the time of delivery, beta cell function as well as beta cell mass return to normal levels. Although to a lesser extent than in rodents, also in humans there have been studies indicating that the beta cell mass may increase during pregnancy and return to normal in the postpartum stage.

When there is no sufficient compensation during pregnancy due to failure in beta cell expansion or function, gestational diabetes mellitus (GDM) occurs.

GDM complicates 2-5% of pregnancies in Caucasian women and is characterized by glucose intolerance with the onset or first diagnosis during pregnancy. GDM can have serious consequences for both the child as well as the mother. Risks to the child include fetal macrosomia as well as long-term health consequences like obesity, hypertension, dyslipidemia, glucose intolerance and type 2 diabetes (T2D). Maternal risks include an increased probability of caesarean delivery accompanied by an increased risk of maternal morbidity.

In women with GDM, glucose homeostasis is returned to normal levels shortly after delivery. However, women with a single gestational diabetes pregnancy present with faster deterioration in insulin sensitivity and beta cell compensation compared to women without a history of gestational diabetes. These women therefore have a 7-fold increased risk of developing T2D in the future. Furthermore, women with a history of GDM have a 10-fold increased risk of developing GDM in future pregnancies.

GDM and T2D The prevalence of T2D in the Netherlands is 600.000-800.000 and each year ~70.000 new patients are diagnosed. Patients with T2D have a 2-4 times increased risk of developing cardiovascular disease. These complications seriously decrease the quality of life and life expectancy of T2D patients. The burden of this disease not only affects these patients but our society as well. Health care costs with respect to diabetes amounted to 814 million euro in 2005 in the Netherlands and indirect costs because of absence of work are unknown but thought to be substantial.

T2D is mainly characterized by defective insulin secretion and peripheral insulin resistance. It develops chronically over years to decades before it becomes apparent. Early in the disease progression, pancreatic beta cells respond to initial insulin resistance by increasing insulin secretion to preserve a near-normal glucose level. Over time the beta cell mass reduces gradually, leading to a decline in insulin secretion causing hyperglycemia. Beta cell failure is dependent on several factors like genetic predisposition, poor dietary control, glucotoxicity and lipotoxicity, liver steatosis and therapy itself.

In the process of development of disease many secondary changes in metabolism, hormonal signaling and body composition occur which are difficult to discriminate from those that initially started the pathophysiological process. Therefore, the early pathogenesis of T2D is still not completely understood. Risk factors for the development of T2D overlap with the risk factors for GDM. These common risk factors suggest an overlapping cause of the disease.

In patients with GDM glucose homeostasis cannot be maintained under conditions of increased metabolic demand. This fact, together with the increased risk of developing T2D in the future suggests a specific predisposition for beta cell dysfunction in these patients.

Beta cell mass in T2D Besides the well-known role of peripheral insulin resistance in the early pathogenesis of T2D, there is also evidence suggesting the importance of beta cell mass. Studies performed on autopsy material of T2D patients in various populations show a significantly reduced beta cell mass. This reduction could be explained by accelerated beta cell death in these patients. A genetic difference in beta cell mass could however also play a role. Large variations in fractional beta cell area have been shown between individuals in the pre- and postnatal growth period. Furthermore, a recent study by Brom et al. suggests that there is a large variation in beta cell mass between individuals. In this study beta cell mass was measured non-invasively in healthy subjects as well as type 1 diabetic patients by 111In-exendin-4 SPECT/CT. While the beta cell mass in these diabetic patients was found to be significantly lower than in healthy subjects, a wide range in beta cell mass was found in both groups. These results are in line with an earlier study where wide ranges in beta cell mass were found in pancreas obtained at autopsy of diabetic and non-diabetic subjects.

An initial deficit in beta cell mass could thus play a key role in the development of T2D. Patients with a history of GDM have a significantly increased risk of developing T2D. While an increase in beta cell mass has been found in healthy women during pregnancy, it is not yet known whether patients with GDM have a deficit in beta cell mass. While little is known about beta cell mass in women with a history of GDM, it is well recognized that these women have a chronic defect in beta cell function that progressively worsens in the years after the pregnancy and mediates their high risk of progression to T2D. This deterioration of beta cell function begins as early as the first year after delivery, is partly driven by hepatic insulin resistance, takes place in the presence of initial normal glucose tolerance, and precedes the development of abnormal glucose tolerance. Accordingly, women with a recent history of GDM represent a patient population in which there is beta cell dysfunction without the potential confounding effect of hyperglycemia (and resultant glucotoxicity).

Evaluation of beta cell mass in women with a history of GDM could thus be very beneficial for our understanding of the role of beta cell mass in the development of T2D. It would be of great interest to examine whether the population of women with a history of gestational diabetes, who have a significantly increased risk of developing T2D, have a lower mean beta cell mass compared to the population of women without a history of gestational diabetes.

Also for the development of new treatment options for T2D, more knowledge on the role of beta cell loss in the development of T2D would be beneficial. While current and new anti-diabetic drugs are mainly targeting insulin secretion and action or glucose uptake, evidence from animal experiments suggests the feasibility of regulating beta cell mass.

Imaging of beta cells in vivo Reliable, sensitive and specific visualization of living pancreatic beta cells in vivo is important to broaden the understanding of the role of beta cell mass in the onset and development of T2D. This could benefit further research in the causes of beta cell failure in T2D and therapeutic options to delay progressive loss of beta cells. Because of the multifactorial nature of T2D disease, defining a study population for assessment of beta cell mass is difficult. Patients with a history of GDM would be a very attractive population to study in this context as an at-risk cohort for T2D. These patients have a clear predisposition for development of T2D evidenced by their increased risk for developing this disease and the faster deterioration of insulin sensitivity and beta cell compensation.

GLP-1 receptor imaging by PET For specific non-invasive imaging of beta cells, investigators have developed a highly beta cell-specific radiolabeled exendin-based GLP-1 (glucagon-like peptide-1) analog which, after radiolabeling, can non-invasively be detected in the human body. GLP-1 is an incretin hormone that specifically binds to beta cells and is responsible for post-prandial insulin-secretion. Its specificity for beta cells has been shown and a linear correlation of the beta cell mass and the signal obtained with this tracer has been established in rats.

GLP-1R imaging has been shown to be suitable for imaging of insulin producing pancreatic neuroendocrine tumours (IPPNET). Furthermore, the feasibility of visualization of transplanted beta cells with GLP-1R imaging has been shown by imaging of autologous islets transplanted into muscle.

ELIGIBILITY:
Inclusion Criteria (women with a history of GDM):

* Pregnancy with diagnosis of GDM, within the last 5 years
* No other previous pregnancies
* Complete resolution of GDM after delivery
* No evidence of T2D at the time of inclusion
* BMI between 17 and 30
* Signed informed consent

Inclusion criteria (women without a history of GDM)

* Pregnancy without problems in glucose homeostasis, within the last 5 years
* No other previous pregnancies
* No evidence of T2D at time of inclusion
* Insulin secretion-sensitivity index-2 (ISSI-2) > 800 on oral glucose tolerance test
* BMI between 17 and 30
* Signed informed consent

Exclusion Criteria:

* Previous treatment (within 6 months) with synthetic exendin
* Breast feeding
* Current pregnancy
* Renal dysfunction
* Liver disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-11-10 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Pancreatic uptake of 68Ga-NODAGA-exendin-4 | 1 year
  Pancreatic tracer uptake by quantitative analysis of PET images

SECONDARY OUTCOMES:
C-peptide, HbA1c | 1 year
  Correlation of tracer uptake and beta cell function

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No